CLINICAL TRIAL: NCT04844554
Title: Protocol of Assistance to Patients With Covid-19 Submitted to Treatment With HD-tDCS: Open Label, Randomized, Controlled Study
Brief Title: Protocol of Assistance to Patients With Covid-19 Submitted to Treatment With HD-tDCS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of Paraíba (Other)
Collaborators: City University of New York (Other); University of Michigan (Other); Rio de Janeiro State University (Other)
Responsible Party: Principal Investigator, Suellen Marinho Andrade, Principal Researcher and Professor, Federal University of Paraíba
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COVID/hd-tDCS
Record Dates: First submitted 2021-03-29; First posted 2021-04-14 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-02

CONDITIONS: Coronavirus; COVID-19 Respiratory Infection
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 - 3.0 mA active HD-tDCS (Experimental): HD-tDCS with 3.0 milliamperes (mA) of intensitive
  Interventions: Other: Active HD-tDCS 3mA
- Group 2 - Sham HD-tDCS (Experimental): Sham HD-tDCS
  Interventions: Other: Sham HD-tDCS

INTERVENTIONS:
Other: Active HD-tDCS 3mA — This group will receive HD-tDCS 3mA intensitie. 0 sessions at ICU simultaneously to physical rehabilitation. The HD- tDCS will be started with a 30 s ramp-up to the desired intensity, which was maintained for 20 min.
  Arms: Group 1 - 3.0 mA active HD-tDCS
Other: Sham HD-tDCS — This group will receive sham HD-tDCS. The intervention will be applied in 10 sessions at ICU simultaneously to physical rehabilitation. The HD- tDCS will be started with a 30 s ramp-up them turn off.
  Arms: Group 2 - Sham HD-tDCS

SUMMARY:
COVID-19 has a variety of symptoms from asymptomatic respiratory dysfunction to death. Considering the pathophysiology of SARS-CoV-2 and its relationship with the neuroimmune system, response, autonomic balance, musculoskeletal and respiratory and neuropsychiatric symptoms presented by patients, the investigators highlight the potential use of non-invasive neuromodulation methods to assess the effectiveness of treating patients with COVID-19, as these techniques can be useful in the management of important clinical aspects in the functional recovery of individuals affected by the disease.

The investigators intend to evaluate the effects of HD- tDCS to promote ventilatory weaning in patients admitted to the Intensive Care Unit (ICU) and to improve the respiratory performance of those hospitalized in nursing beds for treatment of COVID - 19.

ELIGIBILITY:
Intensive Care Unit's Inclusion Criteria:

Patients of at least 18 years-old with a PCR-confirmed SARS-CoV-2 diagnosis and receiving mechanical ventilation at least 48 hours of meeting criteria for moderate to severe acute respiratory distress syndrome (ARDS), under weaning, were enrolled in this study. An ARDS diagnosis was made according to the Berlin Definition criteria.

Intensive Care Unit's Exclusion Criteria:

Patients were excluded if they had a condition that could prevent adequate performance of inspiratory muscle training (e.g., neuropathy or myopathy), pregnancy or active lactation, Richmond Agitation and Sedation Scale (RASS) scores between -2 and + 1, Glasgow Coma Scale (GCS) ≤ 8, consent refusal, and contraindications to brain stimulation (e.g., aneurysm clips).

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-06-20 (Actual); Primary Completion 2022-04-12 (Estimated); Study Completion 2022-10-12 (Estimated)

PRIMARY OUTCOMES:
ICU's primary outcome - number of days alive and free from mechanical ventilation | 28 days
  The primary outcome was ventilator-free days during the first 28 days, defined as the number of days alive and free from mechanical ventilation for at least 48 consecutive hours.

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Paraíba,Department of Psychology, João Pessoa, Paraíba, Brazil